CLINICAL TRIAL: NCT06397833
Title: A Prospective, Observational, Single Centre Study to Assess the Feasibility of the Data Harvested by the Acorai Intracardiac Pressure Monitoring (ICPM) System in Predicting Prognosis in Patients Discharged From Hospital After Treatment for Acute Decompensated Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 334837
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Decompensated Heart Failure
Keywords: heart failure; decompensated heart failure; acorai; artificial intelligence; machine learning generisation; machine learning generization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Decompensated Heart Failure Group: Patient has been admitted to hospital with decompensated heart failure, received at least one dose of an intravenous diuretic, and are awaiting discharge home following their treatment.
  Interventions: Device: Acorai ICPM system

INTERVENTIONS:
Device: Acorai ICPM system — Patient will have the handheld Acorai ICPM system placed on their chest, for a period of 5 minutes for sensor recording time

SUMMARY:
Acorai is developing the Acorai Heart Monitor, a handheld electronic device for monitoring pressures inside the heart in a non-invasive manner, by placing the device on the chest of a patient. Currently these intracardiac pressures are measured in an invasive way, during a right heart catheterisation procedure. This procedure carries risks to the patient. There is a clinical need for a non -invasive, easy to use, tool to monitor patients that suffer from heart failure. The study aim is to use the Acorai device to collect the intracardiac pressure measurements from patients admitted to hospital with heart failure and who are awaiting discharge home. Using the data, we will assess the feasibility of the Acorai derived cardiac output measurements, and assess what data best predicts survival, death, or major adverse cardiac events (MACE)

DETAILED DESCRIPTION:
There is a need for the development of a tool that can help to identify those HF patients at risk of deterioration. The ideal tool would be quick, easy to use, non-invasive, inexpensive and can be performed by any healthcare practitioner or patient themselves (i.e. point of care testing).

The Acorai Heart Monitor device is an extended smartphone case equipped with a combination of microphonic sensors, inertial measurement units, electrocardiographic sensors and photoplethysmography sensor, in a configuration that is designed to enhance low frequency sound and seismic signals pertaining to intracardiac pressure. Each sensor technology has been validated to minimize the risk to the patient. Sensor data is collected to provide clinicians with the patients intracardiac pressures. This is performed by placing the monitoring device on the chest, with a small smart-wrist watch, for a period of five minutes in the supine position. A feasibility study showed Acorai device cardiac output measurements correlate highly with the gold standard right heart catheterisation (RHC) cardiac output measurement.

Intracardiac pressure monitoring is important in HF patients. Studies also show that raised right atrial pressure and pulmonary capillary wedge pressure are predictors of worse outcomes with increased risk of death, cardiovascular hospitalisation or transplantation. Clinicians can only gather intracardiac pressure measurements by undertaking a RHC procedure with fluoroscopy guidance. However, this is an invasive procedure, with radiation exposure, that carries risks including bleeding, stroke, infection and pneumothorax.

This is a prospective, observational, single-site, non-randomised, non-significant risk, single arm, clinical investigation designed to collect non-invasive cardiac output measurements from the Acorai Heart Monitor device The objective of the study is to assess the feasibility of the Acorai ICPM system to predict survival and hospitalisation at 1 year in hospitalised heart failure patients deemed medically fit for discharge.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all the following criteria to be eligible for participation in the clinical investigation

1. Subjects medically fit for discharge following an admission to Hospital with decompensated heart failure requiring intravenous diuretic therapy
2. Subject is willing and physically able to comply with the specified evaluations as per clinical investigation plan, as assessed by the investigator.
3. Subject is able to provide written consent to participate in the study

Exclusion Criteria:

1. Pregnancy
2. Discretionary exclusion when, in the opinion of the investigator, the inclusion of a potential subject is not in their best interest or not in the interest of compliant performance of the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all subjects, over the age of 18 years, who have been admitted to hospital with decompensated heart failure, requiring intravenous diuretic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of the Acorai ICPM system to predict survival and hospitalisation at 1 year in hospitalised heart failure patients deemed medically fit for discharge. | 1 year

SECONDARY OUTCOMES:
To assess the feasibility of the Acorai ICPM system to predict Major adverse cardiac events (MACE) 1 year in hospitalised heart failure patients deemed medically fit for discharge. | 1 year
  MACE includes: acute coronary syndrome (ACS), stroke, cardiovascular related death, heart failure related admission, arrythmia, heart transplantation, mechanical circulatory support
To evaluate which of the measurements provided by the Acorai ICPM system (PASP, mPAP, PADP, mPCWP, mRAP, CO, SV and PVR) best predict prognosis. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Harefield Hospital, Uxbridge, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chahal RS, Chukwu CA, Kalra PR, Kalra PA. Heart failure and acute renal dysfunction in the cardiorenal syndrome. Clin Med (Lond). 2020 Mar;20(2):146-150. doi: 10.7861/clinmed.2019-0422. PMID 32188648
- [Background] Nagai T, Sundaram V, Rothnie K, Quint JK, Shoaib A, Shiraishi Y, Kohsaka S, Piper S, McDonagh TA, Hardman SMC, Goda A, Mizuno A, Kohno T, Rigby AS, Yoshikawa T, Clark AL, Anzai T, Cleland JGF. Mortality after admission for heart failure in the UK compared with Japan. Open Heart. 2018 Sep 11;5(2):e000811. doi: 10.1136/openhrt-2018-000811. eCollection 2018. PMID 30228905
- [Background] Jones NR, Roalfe AK, Adoki I, Hobbs FDR, Taylor CJ. Survival of patients with chronic heart failure in the community: a systematic review and meta-analysis. Eur J Heart Fail. 2019 Nov;21(11):1306-1325. doi: 10.1002/ejhf.1594. Epub 2019 Sep 16. PMID 31523902
- [Background] Mace MI. A Novel Multisensor Device for Absolute Intracardiac Pressure Measurement, Detection, and Management of Heart Failure. JACC Basic Transl Sci. 2023 Apr 24;8(4):377-379. doi: 10.1016/j.jacbts.2023.02.001. eCollection 2023 Apr. No abstract available. PMID 37138811
- [Background] Koehler F, Koehler K, Deckwart O, Prescher S, Wegscheider K, Winkler S, Vettorazzi E, Polze A, Stangl K, Hartmann O, Marx A, Neuhaus P, Scherf M, Kirwan BA, Anker SD. Telemedical Interventional Management in Heart Failure II (TIM-HF2), a randomised, controlled trial investigating the impact of telemedicine on unplanned cardiovascular hospitalisations and mortality in heart failure patients: study design and description of the intervention. Eur J Heart Fail. 2018 Oct;20(10):1485-1493. doi: 10.1002/ejhf.1300. Epub 2018 Sep 19. PMID 30230666
- [Background] Gardner RS, Henderson G, McDonagh TA. The prognostic use of right heart catheterization data in patients with advanced heart failure: how relevant are invasive procedures in the risk stratification of advanced heart failure in the era of neurohormones? J Heart Lung Transplant. 2005 Mar;24(3):303-9. doi: 10.1016/j.healun.2004.01.010. PMID 15737757
- [Background] Ahlgrim C, Kocher S, Minners J, Jander N, Savarese G, Neumann FJ, Arentz T, Jadidi A, Mueller-Edenborn B. Pulmonary Capillary Wedge Pressure during Exercise Is Prognostic for Long-Term Survival in Patients with Symptomatic Heart Failure. J Clin Med. 2022 Oct 6;11(19):5901. doi: 10.3390/jcm11195901. PMID 36233773